CLINICAL TRIAL: NCT06892158
Title: Massage Impact on Sleep in Hospitalization for Pediatric Oncology and Stem Cell Transplant Patients
Brief Title: Massage Impact on Sleep in Pediatric Oncology
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital of Philadelphia (Other)
Collaborators: Massage Therapy Foundation (Other); Children's National Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 24-022048
Record Dates: First submitted 2025-03-18; First posted 2025-03-24 (Actual); Last update posted 2025-03-24 (Actual); Status verified 2025-03

CONDITIONS: Cancer; Pediatric Cancer; Chemotherapy Effect; Acute Myeloid Leukemia; Acute Lymphoblastic Leukemia, Pediatric; Hematopoietic Stem Cell Transplantation (HSCT)
Keywords: Stem cell transplant (SCT); Decreased sleep efficiency; Pediatric cancer diagnosis; Circadian activity rhythm (CAR)
MeSH Terms: conditions — Neoplasms; Leukemia, Myeloid, Acute; Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — Massage; Standard of Care

STUDY DESIGN:
Intervention Model Description: This study is a randomized, two-group design (intervention arm, IA and control arm, CA).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Arm (CA) (Active Comparator): Standard of care.
  Interventions: Other: Standard of care
- Intervention Arm (IA) (Experimental): Massage therapy
  Interventions: Other: Massage therapy

INTERVENTIONS:
Other: Massage therapy — Participants in IA will receive a 20-30-minute massage five days per week for 21 days.
  Arms: Intervention Arm (IA)
Other: Standard of care — Institutional standard of care treatment
  Arms: Control Arm (CA)

SUMMARY:
This study aims to determine the impact of massage therapy for pediatric patients receiving intensive chemotherapy or stem cell transplant (SCT).

DETAILED DESCRIPTION:
Hospitalized pediatric oncology patients report anxiety, pain, disturbed sleep, and excess fatigue. Massage is safe, does not interfere with medications, and has been shown in limited studies to have efficacy in improving sleep as well as decreasing fatigue, anxiety and other symptoms in cancer patients and children with various ailments.

This project aims to determine if individualized massage therapy for hospitalized pediatric patients receiving intensive chemotherapy or stem cell transplant (SCT) is associated with longer duration and improved quality of sleep, more robust circadian rhythms (CARs), improved quality of life (QOL) and reduced fatigue, anxiety, and pain, as compared to a standard of care group.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of cancer, such as acute myeloid leukemia (AML) or relapsed acute lymphoblastic leukemia (rALL) OR admitted to receive autologous or allogeneic HSCT for any indication
2. Expected to be an inpatient for at least 21 days
3. Aged 12 to 21 years at enrollment.
4. Inpatient at Children's National or Children's Hospital of Philadelphia (CHOP).

Exclusion Criteria:

1. Cognitive impairment sufficient to preclude completing questionnaires appropriately
2. Insufficient knowledge of English or Spanish that would prohibit completing the study instruments
3. Previous enrollment

Ages: 12 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 70 (Estimated)
Dates: Start 2025-01-23 (Actual); Primary Completion 2028-01 (Estimated); Study Completion 2028-07 (Estimated)

PRIMARY OUTCOMES:
Improvement in total sleep minutes | 3 weeks
  Change in the total number of sleep minutes over time in the standard of care intervention compared to the change in the total number of sleep minutes over time in the massage therapy intervention. Sleep minutes are measured by actigraphy.

SECONDARY OUTCOMES:
Improvement in sleep quality as demonstrated by circadian activity rhythms (CARs) | 3 weeks
  Amount of dysrgulation in CARs in the standard of care intervention compared to the amount of dysregulation in CARs in the massage therapy intervention. Dysregulation in CARs will be measured by actigraphy (24-h autocorrelation).

CONTACTS AND LOCATIONS:
Overall Officials: Tracey Jubelirer, MD, Principal Investigator — Children's Hospital of Philadelphia
Locations (2):
- United States (2):
  - Children's National Hospital, Washington D.C., District of Columbia
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania